CLINICAL TRIAL: NCT02464995
Title: Bronchial Thermoplasty in Severe Asthma With Frequent Exacerbations
Acronym: THERMASCORT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5886
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Asthma
Keywords: Asthma,; Asthma exacerbation; Bronchial thermoplasty
MeSH Terms: conditions — Asthma | interventions — Bronchial Thermoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thermoplasty group (Experimental): Procedure: Bronchial thermoplasty with the Alair System and conventional therapy
  Interventions: Device: Bronchial thermoplasty with the Alair System
- Control group (No Intervention): Conventional therapy

INTERVENTIONS:
Device: Bronchial thermoplasty with the Alair System
  Arms: Thermoplasty group

SUMMARY:
The purpose of this study is to demonstrate the effectiveness of bronchial thermoplasty in a severe asthmatic population with frequent exacerbations.

This will be a single center randomized and controlled study. Thirty subjects with severe asthma (Gina 4 and 5) with frequent severe exacerbations (four or more bursts of systemic corticosteroids >3 days each in the previous year) will be randomized 1:1 to either the thermoplasty group (bronchial thermoplasty and medical management) or control group (medical management only).

ELIGIBILITY:
Inclusion criteria:

* Age 18-65 years
* Asthma which requires treatment with guidelines suggested medications for GINA steps 4-5
* Four or more bursts of systemic corticosteroids >3 days each in the previous year
* Willingness and ability to give written informed consent

Exclusion criteria:

* Current smoker and former smoker > 10 pack years total smoking history
* Participation in another clinical trial within the prior 4 months
* Omalizumab therapy within the prior 4 months
* Allergic bronchopulmonary aspergillosis
* Patient having had severe exacerbation of their asthma requiring high doses of oral corticosteroids (> 60 mg equivalent prednisolone) more than one month in the previous year
* Post-bronchodilator FEV1 of less than 30%
* Past diagnosis of COPD and chronic respiratory insufficiency
* Known coagulopathy or platelet dysfunction
* Use of anticoagulants
* Use of an internal or external pacemaker or internal cardiac defibrillator
* Contraindication to perform bronchoscopy
* Contraindication to perform general anesthesia
* Significant cardiovascular disease
* Current or recent respiratory tract infection resolved less than 4 weeks
* Known cancer or cancer history less than 12 months
* Pregnancy and nursing mother

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2015-06-09 (Actual); Primary Completion 2020-11-09 (Estimated); Study Completion 2022-11-09 (Estimated)

PRIMARY OUTCOMES:
Severe exacerbation rate (change from baseline) | Baseline, 6 months and 12 months after the last thermoplasty procedure
  A severe exacerbation is defined by a burst of systemic corticosteroids >3 days

SECONDARY OUTCOMES:
Time to the first severe asthma exacerbation | anytime
Mean oral glucocorticosteroid dose (mg equivalent prednisone) | Baseline, 6 and 12 Months
Mild exacerbation rate | Baseline, 6 and 12 Months
Pre- and post-bronchodilator FEV1 | Baseline, 6 and 12 Months
Asthma Control Questionnaire (ACQ) Score | Baseline, 3, 6, 9 and 12 Months
Asthma Quality of Life Questionnaire (AQLQ) Score | Baseline, 3, 6, 9 and 12 Months
Structural airway remodeling using CT | Baseline and 12 Months
Inflammatory cells and markers in induced sputum | Time Frame: Baseline and 12 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France